CLINICAL TRIAL: NCT00144222
Title: A Randomized, Double-Blind Study Comparing a Fixed Dose Combination of Telmisartan 40 mg Plus Hydrochlorothiazide 12.5 mg to Telmisartan 40 mg in Patients Who Fail to Respond Adequately to Treatment With Telmisartan 40 mg
Brief Title: Combination of Telmisartan 40 mg Plus Hydrochlorothiazide (HCTZ) 12.5 mg vs. Telmisartan 40 mg Alone in Patients With Essential Hypertension Who Fail to Respond Adequately to Telmisartan Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.436
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan 40 mg/HCTZ 12.5 mg
Drug: Telmisartan 40 mg

SUMMARY:
The objective of this trial is to demonstrate that the fixed dose combination of telmisartan 40 mg and HCTZ 12.5 mg is superior to the monocomponent of telmisartan (Micardis, Gliosartan, Kinzal, Kinzalmono, Predxal, Pritor, Samertan, Telmisartan) 40 mg in patients with essential hypertension who fail to respond adequately to telmisartan monotherapy.

DETAILED DESCRIPTION:
This is a multi-centre, randomised, double-blind, double-dummy, active-controlled, parallel-group study in patients with essential hypertension who fail to respond adequately to telmisartan (Micardis) 40 mg monotherapy.

After a screening and a 2-week washout period (screening period), the patients will enter 4-week open-label run-in period with telmisartan (Micardis) 40 mg monotherapy to assess eligibility. The study will be terminated for those who have responded to telmisartan (Micardis) 40 mg monotherapy at the end of 4-week open-label run-in period with telmisartan (Micardis) 40 mg monotherapy (mean seated DBP < 90 mmHg). About 200 patients not responding adequately to telmisartan (Micardis) 40 mg monotherapy will be randomised and treated for 8 weeks with once-daily administration of either telmisartan (Micardis) 40 mg or a fixed dose combination of telmisartan 40 mg and HCTZ 12.5 mg (double-blind treatment period).

Study Hypothesis:

The hypothesis is that the fixed dose combination of telmisartan 40 mg and HCTZ 12.5 mg is superior to the monocomponent of telmisartan (Micardis) 40 mg in pat ient with essential hypertension who fail to respond adequately to telmisartan monotherapy.

Comparison(s):

For the primary comparison the change from baseline in mean stated trough DBP at the end of the 8-week double-blind treatment will be expressed.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertensive patients who meet all the criteria as follows:

  * Mean seated DBP must be >= 95 and <= 114 mmHg at Visit 2
  * Mean seated SBP must be >= 140 and <= 200 mmHg at Visit 2
  * Mean seated DBP must be >= 90 and <= 114 mmHg at Visit 3
  * Mean seated SBP must be <= 200 mmHg at Visit 3

Exclusion Criteria:

* Patients taking 4 or more anti-hypertensive medications at Visit 1
* Patients with known or suspected secondary hypertension (renovascular hypertension, primary aldosteronism, pheochromocytoma, etc.)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2005-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08

PRIMARY OUTCOMES:
Change in mean seated trough DBP after eight weeks of the double-blind treatment period | after 8 weeks

SECONDARY OUTCOMES:
Change in seated trough SBP | after 8 weeks
Seated DBP control rate (seated trough DBP < 90 mmHg) | after 8 weeks
Seated DBP response rate V2 (seated trough DBP < 90 mmHg and/or reduction from pseudo-baseline in seated trough DBP ≥ 10 mmHg) | after 8 weeks
Seated DBP response rate V3 (seated trough DBP < 90 mmHg and/or reduction from pseudo-baseline in seated trough DBP ≥ 10 mmHg) | after 8 weeks
Seated SBP response rate V2 (seated trough SBP < 140 mmHg and/or reduction from pseudo-baseline in seated trough SBP ≥ 10 mmHg) | after 8 weeks
Seated SBP response rate V3 (seated trough SBP ≥ 140 mmHg at baseline and seated trough SBP < 140 mmHg and/or reduction from baseline in seated trough SBP ≥ 10 mmHg) | after 8 weeks
Change in trough pulse pressure | after 8 weeks
Plasma concentrations of Telmisartan and HCTZ | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Nippon Boehringer Ingelheim Co., Ltd.
Locations (2):
- Japan (2):
  - Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo